CLINICAL TRIAL: NCT01572402
Title: Postprandial Insulin Secretion, Oxidative Stress and Gastrointestinal Peptides in Patients With Type 2 Diabetes Versus Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Hana Kahleova, Principal Investigator, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 5206
Record Dates: First submitted 2012-04-03; First posted 2012-04-06 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Type 2 Diabetes; Postprandial Oxidative Stress
Keywords: Diet; Gastrointestinal peptides; Insulin secretion; Oxidative stress; Plasma lipids; Postprandial; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with type 2 diabetes (Experimental): Study group: 40 individuals with type 2 diabetes treated by diet and/or oral hypogylycemic agents, diabetes duration at least 1 year, both men and women, age 30-65 years, BMI 27-50 kg/m². The subjects will be explained aims, methods and risks of the study and they will sign informed consent
  Interventions: Other: Bagueutte Cheese Gourmet (Crocodille); Other: Cous-cous sandwich; Other: McCountry sandwich (McDonald's)
- Healthy subjects (Active Comparator): Mean and women, age 30-70 years, no diabetes, no metabolic syndrome
  Interventions: Other: Bagueutte Cheese Gourmet (Crocodille); Other: Cous-cous sandwich; Other: McCountry sandwich (McDonald's)

INTERVENTIONS:
Other: Bagueutte Cheese Gourmet (Crocodille) — 180g, energy 452.8 Kcal/1895.7 kJ, composition: carbohydrates 49,2 g (44,55%), proteins 18,5 g (16,74%), lipids 18,8 g (38,7%), of which saturated 6,8 g, monounsaturated 6,0 g, polyunsaturated 5,0 g.
Other: Cous-cous sandwich — 235 g, energy 455,88 Kcal /1907,4 kJ, composition: carbohydrates 59,54 g (52,24%), proteins 12,47 g (10,57% %), lipids 18,85 g (37,31%), of which saturated 6,2 g, monounsaturated 11,49 g, polyunsaturated 28,26 g
Other: McCountry sandwich (McDonald's) — 150g, 455 kcal/1903,72 kJ, composition: carbohydrates 31 g (27,25%), proteins 24 g (21,1%), lipids 26 g (51,43%), of which saturated 10 g (38,45%)

SUMMARY:
Insulin secretion, plasma lipids, oxidative stress markers and gastrointestinal peptides will be measured in patients with type 2 diabetes versus healthy subjects in a fasting status and in response to standard meals (at times 0', 30', 60', 120' and 180').

ELIGIBILITY:
Inclusion Criteria:

* 40 individuals with type 2 diabetes treated by diet only or oral hypogylycemic agents,
* diabetes duration at least 1 year,
* both men and women,
* age 30-65 years,
* BMI 27-50 kg/m². The subjects will be explained aims, methods and risks of the study and they will sign informed consent

Exclusion Criteria:

* gravidity,
* lactation,
* drug abuse,
* insulin therapy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Postprandial oxidative stress | up to 2 months
Postprandial plasma concentrations of gastrointestinal peptides | up to 2 months

SECONDARY OUTCOMES:
Postprandial insulin secretion - relationship to oxidative stress and gastrointestinal peptides | up to 2 months
Postprandial plasma lipids | up to 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hana Kahleova, Prague, Czechia

REFERENCES:
- [Derived] Belinova L, Kahleova H, Malinska H, Topolcan O, Vrzalova J, Oliyarnyk O, Kazdova L, Hill M, Pelikanova T. Differential acute postprandial effects of processed meat and isocaloric vegan meals on the gastrointestinal hormone response in subjects suffering from type 2 diabetes and healthy controls: a randomized crossover study. PLoS One. 2014 Sep 15;9(9):e107561. doi: 10.1371/journal.pone.0107561. eCollection 2014. PMID 25222490
- [Derived] Malinska H, Kahleova H, Topolcan O, Vrzalova J, Oliyarnyk O, Kazdova L, Belinova L, Hill M, Pelikanova T. Postprandial oxidative stress and gastrointestinal hormones: is there a link? PLoS One. 2014 Aug 20;9(8):e103565. doi: 10.1371/journal.pone.0103565. eCollection 2014. PMID 25141237